CLINICAL TRIAL: NCT03419312
Title: Cerebral PET Patterns, Inflammatory Biomarkers and Outcome in Patients Treated With Burst Spinal Cord Stimulation for Chronic Low Back and Leg Pain: A Randomized Controlled Clinical Trial
Brief Title: PET Patterns, Biomarkers and Outcome in Burst SCS Treated FBSS Patients
Acronym: PET-SCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uppsala University (Other)
Collaborators: Linkoeping University (Other Government); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB 2017/110/1
Record Dates: First submitted 2017-11-27; First posted 2018-02-01 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: FBSS; Pain, Intractable; Low Back Pain; Radicular; Neuropathic, Lumbar, Lumbosacral
Keywords: Spinal Cord Stimulation; Burst Spinal Cord Stimulation; SCS
MeSH Terms: conditions — Pain, Intractable; Low Back Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: Patients are randomized to 1 of 2 different treatment sequences:
  Sequence A: Active burst stimulation followed by sham stimulation. Sequence B: Sham stimulation followed by burst stimulation. Sham and burst stimulation are separated by 7 days washout.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The stimulation periods with sham stimulation and burst are blinded to all included in the study except SCS nurse 1 who program and reset IPG during study phase 2.
  Sham stimulation is achieved by switching of the stimulation equipment in connection with programming prior to the start of the current stimulation period. The programming procedure is identical before burst and sham stimulation periods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study sequence A (Experimental): Proclaim™ Elite 5: Burst - Washout - Sham
  1. 14 days of burst stimulation.
  2. 7 days washout.
  3. 14 days of sham stimulation.
  Interventions: Device: Proclaim™ Elite 5: Burst - Washout - Sham
- Study sequence B (Experimental): Proclaim™ Elite 5: Sham - Washout - Burst
  1. 14 days of sham stimulation.
  2. 7 days washout.
  3. 14 days of burst stimulation.
  Interventions: Device: Proclaim™ Elite 5: Sham - Washout - Burst

INTERVENTIONS:
Device: Proclaim™ Elite 5: Burst - Washout - Sham — All implanted hardware manufactured by S:t Jude Medical/Abbot:
  Implantable Pulse Generator (IPG): Proclaim™ Elite 5 IPG, model 3660. Electrode: Octrode percutaneous lead, 60 cm, model 3161. Anchor: Long lead anchor, model 1106.
  Other Names: Burst DR; Spinal Cord Stimulation
  Arms: Study sequence A
Device: Proclaim™ Elite 5: Sham - Washout - Burst — All implanted hardware manufactured by S:t Jude Medical/Abbot:
  Implantable Pulse Generator (IPG): Proclaim™ Elite 5 IPG, model 3660. Electrode: Octrode percutaneous lead, 60 cm, model 3161. Anchor: Long lead anchor, model 1106.
  Other Names: Burst DR; Spinal Cord Stimulation
  Arms: Study sequence B

SUMMARY:
The primary aim of this study is to investigate cerebral mechanisms of burst stimulation in Failed Back Surgery Syndrome (FBSS) patients treated with Burst Spinal Cord Stimulation (SCS) for chronic back and leg pain. This study is a single center, prospective, blinded, randomized crossover trial with two 14 days treatment periods and two treatment arms (burst before sham stimulation or sham before burst stimulation).

DETAILED DESCRIPTION:
Background and rationale:

Tonic spinal cord stimulation for chronic primarily neuropathic pain har been used for over 50 years. Tonic stimulation in frequencies from 20 to 70 Hz produces analgesia and paresthesia in the targeted area.

Burst stimulation, a novel spinal cord stimulation pattern, is an intermittent high frequency parenthesis-free therapy. This stimulation pattern consist of 5 spikes with an inter-spike frequency of 500 Hz, delivered at 40 Hz.

Clinical effectiveness and noninferiority of Burst stimulation has been proved. A few studies suggest that Burst stimulation induce different activities in cerebral pathways, compared with tonic stimulation. Patient reported attention to pain assessed by the pain vigilance and awareness questionnaire (PVAQ) seems to differ between burst and tonic spinal cord stimulation. This trial is designed to investigate cerebral mechanisms of burst stimulation, using PET O15-water measured blood flow and tissue perfusion as a proxy for cerebral activity.

Key events in study implementation:

Study phase 1

* Study Inclusion and baseline visit.
* Implantation of spinal cord stimulation system.

Study phase 2:

* Study visit 1(study day 0): Collection of Patient Reported Outcome Measurements (PROM) data, Randomization to study sequence, blood sampling, PET 0, programming of SCS-system.
* Study visit 2 (study day 14): Blood sampling, PET 1, collection of PROM-data, SCS system switched off for washout.
* Study visit 3 (study day 21): Collection of PROM-data, programming of SCS-system, blood sampling.
* Study visit 4 (study day 35): Blood sampling, PET 2, collection of PROM-data, programming of SCS-system.

ELIGIBILITY:
Inclusion Criteria:

1. Occurrence of chronic pain in the lumbosacral region, as well as unilateral or bilateral leg pain.
2. Prior lumbar surgery in medical history.
3. Diagnosed with neuropathic pain in the lower extremities and graded as probable neuropathic pain or definite neuropathic pain according International Association for the Study of Pain (IASP) criteria.
4. Patient report largely unchanged pain condition last 6 months.
5. Patient has undergone a 7 day SCS trial with epidural burst stimulation with the following results:

   1. At least 75% coverage of the painful area of tonic stimulation before start of burst trial stimulation.
   2. At least 50% reduction in pain intensity, measured via BPI, item 5 from baseline of trial to end of trial period.
6. The patient is ≥ 18 years of age and < 60 years of age.
7. The patient must willingly participate in all parts of the study, as well as having the ability to complete the entire study plan.
8. Patient must certify that he / she understands the study plan, as well as voluntarily sign informed consent to participate in the study.
9. Must be able to sit still for a minimum of 45 minutes and be able to follow restrictions related to the PET survey.

Exclusion Criteria:

1. The patient has other current pain conditions than back and leg pain after back surgery.
2. The patient is treated with opioids exceeding 80 milligrams of Morphine per day or is considered at risk for development of problematic opioid use.
3. The patient suffers from an untreated depression or anxiety.
4. The patient can not complete the study plan.
5. The patient is unable to read or write Swedish.
6. The patient is currently participates in another clinical trial.
7. A history of previous PET scan or other substantial radiation dose in the last 5 years.
8. The patients is suffering from claustrophobia.
9. Ongoing pregnancy or planned pregnancy during study time.
10. The patient has contraindications for arterial catheterization.
11. The patient is previously treated with spinal cord stimulation.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 6 female and 6 male subjects will be included.
Enrollment: 12 (Estimated)
Dates: Start 2018-02-11 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change in regional cerebral blood flow measured with 15O-water Positron Emission. Tomography (PET) | PET is performed at study day 0 (baseline), day 14 and day 35.
  35 Volume of Interest (VOI) will be applied to each PET scan using the PVElab software. Cerebral blood flow (CBF) and perfusable tissue fraction (PTF) will be calculated for each VOI at each scan. Same tests will be done at voxel level with the Statistical Parameter Mapping Software (SPM12), to identify areas with changed CBF or PTF that do not correspond to VOI in the template.

SECONDARY OUTCOMES:
Semiquantitative assessment of protein levels associated with inflammation. | Measured at day 0 (baseline), day 14, day 21 and day 35.
  Level of normalized protein expression (NPX) in plasma, assessed by a multiplex proximity extension assay panel (Olink Bioscience, Uppsala, Sweden).
Back and leg pain | Measured at visit day 0 (baseline), day 14 and day 35.
  Measured using a 100mm Visual Analog Scale (VAS) for back and leg pain, respectively. Scale range: 0 mm indicates no pain (minimum), 100 mm indicates worst imaginable pain (maximum).
General pain | Measured at day 0 (baseline), day 14 and day 35.
  General pain measured by Brief Pain Inventory (BPI) item 3, 4, 5 and 6
Pain inference | Measured at day 0 (baseline), day 14 and day 35.
  Measured by BPI item 9A-9G
Disability | Measured at day 0 (baseline), day 14 and day 35.
  Disability measured by Oswestry Disability Index (ODI).
Pain Catastrophizing | Measured at day 0 (baseline), day 14 and day 35.
  Measured by Pain Catastrophizing Scale (PCS).
Pain Vigilance and Awareness | Measured at day 0 (baseline), day 14 and day 35.
  Measured by the Pain Vigilance and Awareness Questionnaire (PVAQ).
Global Impression of Change | Measured at day 14 and day 35.
  Impression of change in health status assessed by the inventory Patient Global Impression of Change (PGIC).
Depression | Measured at day 0 (baseline), day 14 and day 35.
  Symptoms of depression is assessed by the inventory Patient Health Questionnaire (PHQ-9).
Anxiety | Measured at day 0 (baseline), day 14 and day 35.
  Symptoms of anxiety is assessed by the inventory Generalized Anxiety Disorder Screener (GAD-7).

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Karlsten, MD, PhD, Principal Investigator — rolf.karlsten@akademiska.se
Locations (1):
- Uppsala University Hospital, Uppsala University, Dept. of Surgical Sciences and Dept. of Medicinal Chemistry, Div. of Molecular Imaging., Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473